CLINICAL TRIAL: NCT00586300
Title: Multidimensional Intervention in Early Osteoarthritis (The Knee Study)
Brief Title: Community-Based Programs for Improving Physical Function in People With Early Knee Osteoarthritis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Arizona (Other)
Collaborators: National Institute of Arthritis and Musculoskeletal and Skin Diseases (NIAMS) (NIH)
Responsible Party: Principal Investigator, Scott Going, Principal Investigator, University of Arizona
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: R01AR047595 (NIH); R01AR047595 (NIH)
Record Dates: First submitted 2007-12-28; First posted 2008-01-04 (Estimated); Last update posted 2012-06-21 (Estimated); Status verified 2012-06

CONDITIONS: Osteoarthritis
Keywords: Knee pain
MeSH Terms: conditions — Osteoarthritis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 (Active Comparator): Physical training program
  Interventions: Other: Physical training program
- 2 (Active Comparator): Self-management training program
  Interventions: Behavioral: Self-management training program
- 3 (Active Comparator): Physical and self-management training programs
  Interventions: Other: Physical training and self-management training programs

INTERVENTIONS:
Other: Physical training program — The physical training will be completed in two phases. In Phase 1, which will last 9 months, participants will complete the program under the supervision of an experienced trainer. Sessions will occur three times each week in a designated study facility. The program will include the following components: stretching and balance, flexibility and range of motion, muscle strengthening, and aerobics. The program will also emphasize the importance of individualizing exercise regimens according to each person's specific needs (function and fitness). In Phase 2, the primary objective will be to promote long-term exercise (for up to 24 months from the time of study entry) that incorporates the four modalities of exercise instruction introduced in Phase 1, but on an independent basis.
  Other Names: Exercise group
  Arms: 1
Behavioral: Self-management training program — The self-management training program is designed to target primarily coping skills and self-efficacy. This will be accomplished by using a variety of educational and behavioral methods. The program will be delivered in two phases. The initial 9-month phase will consist of 12 weekly 60-minute classroom sessions, followed by 24 weeks of a structured telephone intervention program. Phase 2 will continue to incorporate the telephone intervention program, at less frequent intervals, for up to 24 months from the time of study entry.
  Arms: 2
Other: Physical training and self-management training programs — This "multidimensional" intervention will combine both the physical training and self-management training programs described for Groups 1 and 2.
  Other Names: Combo Group
  Arms: 3

SUMMARY:
Osteoarthritis (OA) is the most common joint-related disease and most prevalent form of arthritis in the United States. Pain relievers and anti-inflammatory medications are the most commonly prescribed treatments for OA. These medications, however, cannot completely alleviate OA symptoms. Additional recommended strategies for managing OA include physical and occupational therapy, exercise, and patient education. This study will compare the effectiveness of a physical training program, a self-management training program, and a program including both physical and self-management training for improving physical function in people with early stage knee OA.

DETAILED DESCRIPTION:
There is no cure for arthritis; therefore, it is important to develop treatments to effectively manage the disease. The primary goals of arthritis management are to reduce pain and improve functional ability and quality of life. Existing treatments, including pain relievers and anti-inflammatory medications, can only partially manage OA symptoms. Few studies, however, have been conducted to evaluate complementary measures, such as exercise and education. This study will compare a physical training program, a self-management training program, and a program including both physical and self-management training to determine their effectiveness in improving physical function in people with early stage knee OA.

Participants in this 2-year study will first undergo a physical evaluation that will include answering a questionnaire and having knee x-rays. Participants will then be randomly assigned to one of three treatment groups. All three treatments will include a 9-month supervised phase (Phase 1) and a 15-month maintenance phase (Phase 2).

* Group 1 participants will partake in a community-based arthritis self-management program. Phase 1 will include weekly 75-minute training sessions for 3 months. These sessions will be led by healthcare professionals and will address topics about arthritis and its treatment, healthy lifestyle, and physical activity. After completing the training sessions, participants will be contacted weekly by telephone for 3 months to discuss their progress. Then the telephone contacts will occur once every other week for the next 3 months. During Phase 2 of the self-management training program, participants will continue to receive telephone contacts from the project team to help support and promote the skills introduced during the training sessions. These contacts will occur monthly for 3 months and then every other month for the remainder of the study.
* Group 2 participants will first attend an orientation workshop and then start a long-term physical training program that will include components of balance, flexibility, muscle strengthening, and aerobic conditioning. During Phase 1, participants will attend three physical training sessions per week. During Phase 2, participants will have the option to continue the program in the location of their choice. Study staff will contact participants monthly by phone to discuss their progress. Participants may meet with the trainer on an as-needed basis for additional assistance with the program. They will also keep a log to track attendance and progress, and they will mail in the log monthly.
* Group 3 participants will complete both the physical and self-management training programs and will follow the schedules outlined for Groups 1 and 2.

All participants will complete questionnaires before beginning their assigned training programs and then every 3 months till Month 24. The questionnaires will take between 30 and 60 minutes to complete. At various times during the study, participants will measure their activity levels with a pedometer or an accelerometer. Prior to starting the training programs, at Month 9, and after completing the training programs, participants will complete several tests to measure their physical capabilities and muscle strength. Upon completing the training programs, participants will receive a follow-up x-ray of their knees at an assigned radiology clinic. They will also be asked to provide feedback on their study experiences via a mailer questionnaire, and they may be asked to provide feedback in a short telephone interview.

ELIGIBILITY:
Inclusion criteria:

* History of pain on most days (i.e., 4 or more days in a week) in one or both knees for at least 4 months during the year prior to study entry
* Duration of symptoms (defined as pain on most days for at least 4 months in 1 year) of less than 5 years
* Radiographic evidence of grade II knee OA
* Some level of disability, represented as a score of 3 or higher for at least three of the following WOMAC Index items: descending or ascending stairs; walking; bending; and performing daily activities

Exclusion criteria:

* Any uncontrolled medical condition that could prevent safe participation in the study (e.g., uncontrolled heart disease, blood pressure, or respiratory conditions)
* Any neurological condition that could affect coordination
* Inflammatory arthritis (e.g., rheumatoid or psoriatic arthritis)
* Participates in aerobic activity or resistance training for more than 60 minutes per week
* History of knee surgery
* Radiographic grade I, III-IV (Kellgren and Lawrence classification)
* Body mass index of at most 37.5 Kg/m2 (Individuals over this limit will be advised to follow a weight loss program and achieve stable weight for 6 months prior to participation.)
* History of a knee corticosteroid injection in the 3 months prior to study entry
* Plans to move from the local area
* Plans to become pregnant during the study

Ages: 35 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 294 (Actual)
Dates: Start 2003-06; Primary Completion 2009-05 (Actual); Study Completion 2009-05 (Actual)

PRIMARY OUTCOMES:
Knee function, as measured by the ERGOS machine | Measured at baseline and Months 9 and 24

SECONDARY OUTCOMES:
Pain, as measured by the visual analogue scale (VAS) and the Pain Subscale of the Western Ontario and MacMasters Universities (WOMAC) | Measured at baseline and Months 3, 9, 18, and 24
Coping efficacy, self-efficacy, and health-related quality of life, as measured by the Client Satisfaction Questionnaire (CSQ) | Measured at baseline and Months 3, 9, 18, and 24
Arthritis self-efficacy scale | Measured at baseline and Months 3, 9, 18, and 24
Positive and Negative Affect Schedule (PANAS) | Measured at baseline and Months 3, 9, 18, and 24
SF-36 Health Survey | Measured at baseline and Months 3, 9, 18, and 24
EuroQuol | Measured at baseline and Months 3, 9, 18, and 24
Medical Outcomes Social Support Survey | Measured at baseline and Months 3, 9, 18, and 24

CONTACTS AND LOCATIONS:
Overall Officials: Scott B. Going, PhD, Principal Investigator — University of Arizona
Locations (1):
- University of Arizona, Tucson, Arizona, United States

REFERENCES:
- [Result] Wright LJ, Zautra AJ, Going S. Adaptation to early knee osteoarthritis: the role of risk, resilience, and disease severity on pain and physical functioning. Ann Behav Med. 2008 Aug;36(1):70-80. doi: 10.1007/s12160-008-9048-5. Epub 2008 Aug 21. PMID 18716855
- [Derived] McKnight PE, Kasle S, Going S, Villanueva I, Cornett M, Farr J, Wright J, Streeter C, Zautra A. A comparison of strength training, self-management, and the combination for early osteoarthritis of the knee. Arthritis Care Res (Hoboken). 2010 Jan 15;62(1):45-53. doi: 10.1002/acr.20013. PMID 20191490
- [Derived] Farr JN, Going SB, McKnight PE, Kasle S, Cussler EC, Cornett M. Progressive resistance training improves overall physical activity levels in patients with early osteoarthritis of the knee: a randomized controlled trial. Phys Ther. 2010 Mar;90(3):356-66. doi: 10.2522/ptj.20090041. Epub 2010 Jan 7. PMID 20056719
- [Derived] Farr JN, Going SB, Lohman TG, Rankin L, Kasle S, Cornett M, Cussler E. Physical activity levels in patients with early knee osteoarthritis measured by accelerometry. Arthritis Rheum. 2008 Sep 15;59(9):1229-36. doi: 10.1002/art.24007. PMID 18759320
- See also: Click here for more information about the Knee Study — http://www.arthritis.arizona.edu